CLINICAL TRIAL: NCT00925899
Title: Melatonin for Fatigue and Other Symptoms in Patients With Advanced Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: I.M Daehnfeldt Foundation (Unknown); Danish Cancer Society (Other); Aase and Ejnar Danielsens Foundation (Other); Beckett Foundation (Other); The Andersen-Isted Foundation (Unknown)
Responsible Party: Principal Investigator, Lise Pedersen, MD, DMSc, Bispebjerg Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Feldt-01
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-03

CONDITIONS: Cancer; Fatigue
Keywords: Melatonin; Palliative care; Advanced cancer; Symptoms; Quality of life; Randomized controlled trial
MeSH Terms: conditions — Neoplasms; Fatigue | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melatonin (Experimental): 20 mg
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — 20 mg melatonin orally every evening about 1 hour before bedtime for one week. After having participated in the cross-over part of the trial (one week of melatonin followed by one week of placebo, or the other way around), the participant may receive melatonin for 6 weeks.
  Arms: Melatonin
Drug: Placebo — Placebo tablet orally every evening about one hour before bedtime for one week. After having participated in the cross-over part of the trial (one week of placebo followed by one week of melatonin, or the other way around), the participant may receive melatonin for 6 weeks.
  Arms: Placebo

SUMMARY:
BACKGROUND:

Patients with advanced cancer often suffer from fatigue and other symptoms and problems such as insomnia, appetite loss and pain. Problems that may have great consequences for their quality of life. Several studies suggest that a supplement of the hormone melatonin (MLT) may have a beneficial effect on these symptoms/problems. This needs further investigation.

AIM:

To investigate if a supplement of melatonin have an effect on a) fatigue (the primary outcome of the trial), b) the symptoms insomnia, appetite loss, depression and pain, and c) overall quality of life.

METHODS AND PATIENTS:

The trial takes place in the Department of Palliative Medicine, Bispebjerg Hospital, and 50 patients will participate. The participants have to be 18 years or above, have advanced cancer, and suffer from quite a bit or very much fatigue.

The study consists of two parts. In part I it is investigated if melatonin has a better effect than placebo on the outcomes mentioned above. This part is a consecutive, prospective, double blinded, randomized (MLT vs. placebo), cross-over study where the patients serve as their own control. In part II the effect of melatonin over time is investigated. Part II is a consecutive, prospective, open-label study.

The outcomes are assessed with weekly questionnaires (MFI-20 and EORTC QLQ-C15PAL) and a few daily diary questions.

Melatonin has been used in several studies, and the general conclusion is that it is a safe substance with few adverse drug reactions.

PERSPECTIVES:

If melatonin has the potential to alleviate fatigue and other symptoms in patients with advanced cancer and enhance the quality of life of these patients, this will be of benefit to many future patients. Trials such as this are important both nationally and internationally to develop an evidence-based palliative medicine.

ELIGIBILITY:
Inclusion Criteria:

* Answered "quite a bit" or "very much" to the question "were you tired?" (from EORTC QLQ-C15-PAL)
* Cancer in a palliative phase
* Written informed consent
* Age 18 years or above

Exclusion Criteria:

* Not capable of understanding or judging information, or fill out a questionnaire
* Untreated anemia (Hb <= 6,0 mmol/L)
* Untreated hypocalcaemia
* Systolic blood pressure < 100
* In treatment with coumadin
* Receiving unstable doses of methylphenidate, corticosteroids or sleeping medicine the past two weeks
* TSH < 0.50 or > 5.50 mcL/mL
* Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lise Pedersen, MD, DMSc., Principal Investigator — Department of Palliative Medicine, Bispebjerg Hospital
Locations (1):
- Department of Palliative Medicine, Bispebjerg Hospital, Copenhagen, Denmark

REFERENCES:
- [Result] Lund Rasmussen C, Klee Olsen M, Thit Johnsen A, Petersen MA, Lindholm H, Andersen L, Villadsen B, Groenvold M, Pedersen L. Effects of melatonin on physical fatigue and other symptoms in patients with advanced cancer receiving palliative care: A double-blind placebo-controlled crossover trial. Cancer. 2015 Oct 15;121(20):3727-36. doi: 10.1002/cncr.29563. Epub 2015 Jul 15. PMID 26178160

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 72 patients were randomised in the study. 50 patients completed the first part of the stud, only 44 patients were complete compliers (having taking their melatonin and placebo for at least five days each week and having answered the questionnaires at all times). The primary analysis is of the 44 complete compliers.
Groups:
- Part 1: Melatonin, Then Placebo: First one week Melatonin: 20 mg melatonin orally every evening about 1 hour before bedtime for one week.
  Then one week Placebo: Placebo tablet orally every evening about one hour before bedtime for one week.
- Part 1: Placebo, Then Melatonin: First one week Placebo: Placebo tablet orally every evening about one hour before bedtime for one week.
  Then one week Melatonin: 20 mg melatonin orally every evening about 1 hour before bedtime for one week.
Period: Part 1
Arm/Group | Part 1: Melatonin, Then Placebo | Part 1: Placebo, Then Melatonin
Started | 34 | 38
Completed | 23 | 27
Not Completed | 11 | 11
Not completed — Death | 1 | 2
Not completed — Withdrawal by Subject | 10 | 9
Period: Part 2
Arm/Group | Part 1: Melatonin, Then Placebo | Part 1: Placebo, Then Melatonin
Started (Nine patients withdrew before part two because they did not wish to continue in the study) | 15 (All patients received the same intervention in the second part of the study (20 mg melatonin)) | 21 (Nine patients withdrew because they did not wish to continue in the study)
Completed | 9 | 9
Not Completed | 6 | 12

BASELINE CHARACTERISTICS:
Groups:
- Melatonin, Then Placebo: Melatonin then placebo: 20 mg melatonin orally every evening about 1 hour before bedtime for one week. Then 1 week placebo.
- Placebo. Then Melatonin: Placebo then melatonin: Placebo tablet orally every evening about one hour before bedtime for one week. Then one week melatonin 20 mg orally.
- Total: Total of all reporting groups
Arm/Group | Melatonin, Then Placebo | Placebo. Then Melatonin | Total
Number analyzed (Participants) | 34 | 38 | 72
Age, Continuous [Mean (Full Range); unit: years] | 65 [35 to 84] | 62 [33 to 89] | 63 [33 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 49
  Male | 10 | 13 | 23

OUTCOME MEASURES:

1. Primary Outcome: Fatigue as Measured by the Physical Fatigue Scale in the The Multidimensional Fatigue Inventory (MFI) (Smets EM, Garssen B, Bonke B, et al., J Psychosom Res 39:315-325, 1995)
Description: Primary outcome: Change from baseline to week one in intervention group minus change from baseline to week one in control group.
  Because it was a cross-over trial this was calculated the following way:
  Outcomes for arm 1 (melatonin then placebo) were calculated as the difference in mean change scores between week 1 and week 2 (scores for day 7 to day 1-scores for day 17 to day 10). Outcomes for arm 2 (placebo then melatonin) were calculated as the difference in mean change scores between week 2 and week 1 (scores for day 17 to day 10-scores for day 7 to day 1).
  The physical fatigue scale conists of four item each ranging from one to five. The four item were summed and the scae was converted to 0 to 100, where 100 indicated maximum fatigue.
Time Frame: One week
Population: The primary analysis was a per protocol analysis including only complete compliers, defined as those patients who had consumed at least 5 capsules per week for the 2 weeks in part 1 and who had answered the MFI-20 on days 1, 7, 10, and 17.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Melatonin Then Placebo: 20 mg Melatonin orally every evening about 1 hour before bedtime for one week. Then Placebo tablet orally every evening about one hour before bedtime for one week. Three days wash out in between.
- Placebo Then Melatonin: Placebo tablet orally every evening about one hour before bedtime for one week. Then melatonin 20 mg melatonin orally every evening about 1 hour before bedtime for one week. Three days wash out in between.
Arm/Group | Melatonin Then Placebo | Placebo Then Melatonin
Number analyzed (Participants) | 21 | 23
units on a scale | -1.1 (15.9) | -3.9 (18.1)

2. Secondary Outcome: Insomnia Measured by the Insomnia Item in the Questionnaire EORTC QLQ-C15-PAL
Description: Primary outcome: Change from baseline to week one in intervention group minus change from baseline to week one in control group.
  Because it was a cross-over trial this was calculated the following way:
  Outcomes for arm 1 (melatonin then placebo) were calculated as the difference in mean change scores between week 1 and week 2 (scores for day 7 to day 1-scores for day 17 to day 10). Outcomes for arm 2 (placebo then melatonin) were calculated as the difference in mean change scores between week 2 and week 1 (scores for day 17 to day 10-scores for day 7 to day 1).
  Insomnia was converted to a 0 til 100 scale according to the scoring manual for EORTC QLQ C15-PAL where 100 indicated maximum insomnia.
Time Frame: One week
Population: Complete compliers
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Melatonin Then Placebo | Placebo Then Melatonin
Number analyzed (Participants) | 21 | 23
units on a scale | -9.9 (23.4) | -4.6 (30.9)

3. Secondary Outcome: Emotional Function as Measured by the Questionnaire EORTC QLQ-C15-PAL (Groenvold M, Petersen MA, Aaronson NK, et al, Eur J Cancer 42:55-64, 2006)
Description: Change from baseline to week one in intervention group minus change from baseline to week one in control group.
  Because it was a cross-over trial this was calculated the following way:
  Outcomes for arm 1 (melatonin then placebo) were calculated as the difference in mean change scores between week 1 and week 2 (scores for day 7 to day 1-scores for day 17 to day 10). Outcomes for arm 2 (placebo then melatonin) were calculated as the difference in mean change scores between week 2 and week 1 (scores for day 17 to day 10-scores for day 7 to day 1).
  Emotional function was converted to a 0 til 100 scale according to the scoring manual for EORTC QLQ C15-PAL where 100 indicated the best possible emotional function.
  Note outcome reported for complete compliers
Time Frame: One week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Melatonin Then Placebo | Placebo Then Melatonin
Number analyzed (Participants) | 21 | 23
units on a scale | -0.6 (23.5) | 3.3 (18.5)

4. Secondary Outcome: Pain as Measured by the Questionnaire EORTC QLQ-C15-PAL (Groenvold M, Petersen MA, Aaronson NK, et al, Eur J Cancer 42:55-64, 2006)
Description: Change from baseline to week one in intervention group minus change from baseline to week one in control group.
  Because it was a cross-over trial this was calculated the following way:
  Outcomes for arm 1 (melatonin then placebo) were calculated as the difference in mean change scores between week 1 and week 2 (scores for day 7 to day 1-scores for day 17 to day 10). Outcomes for arm 2 (placebo then melatonin) were calculated as the difference in mean change scores between week 2 and week 1 (scores for day 17 to day 10-scores for day 7 to day 1).
  Pain was converted to a 0 til 100 scale according to the scoring manual for EORTC QLQ C15-PAL where 100 indicated maximum pain.
  Note outcome reported for complete compliers
Time Frame: One week
Population: Complete compliers
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Melatonin Then Placebo | Placebo Then Melatonin
Number analyzed (Participants) | 21 | 23
units on a scale | 0.8 (19.3) | 1.9 (22.2)

5. Secondary Outcome: Quality of Life as Measured by the Questionnaire EORTC QLQ-C15-PAL (Groenvold M, Petersen MA, Aaronson NK, et al, Eur J Cancer 42:55-64, 2006)
Description: Change from baseline to week one in intervention group minus change from baseline to week one in control group.
  Because it was a cross-over trial this was calculated the following way:
  Outcomes for arm 1 (melatonin then placebo) were calculated as the difference in mean change scores between week 1 and week 2 (scores for day 7 to day 1-scores for day 17 to day 10). Outcomes for arm 2 (placebo then melatonin) were calculated as the difference in mean change scores between week 2 and week 1 (scores for day 17 to day 10-scores for day 7 to day 1).
  Quality of Life was converted to a 0 til 100 scale according to the scoring manual for EORTC QLQ C15-PAL where 100 indicated best possible quality of life.
  Note outcome reported for complete compliers
Time Frame: One week
Population: Complete compliers
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Melatonin Then Placebo | Placebo Then Melatonin
Number analyzed (Participants) | 21 | 23
units on a scale | -0.8 (13.6) | -3.2 (19.2)

6. Secondary Outcome: Appetite Loss as Measured by the Questionnaire EORTC QLQ-C15-PAL (Groenvold M, Petersen MA, Aaronson NK, et al, Eur J Cancer 42:55-64, 2006)
Description: Change from baseline to week one in intervention group minus change from baseline to week one in control group.
  Because it was a cross-over trial this was calculated the following way:
  Outcomes for arm 1 (melatonin then placebo) were calculated as the difference in mean change scores between week 1 and week 2 (scores for day 7 to day 1-scores for day 17 to day 10). Outcomes for arm 2 (placebo then melatonin) were calculated as the difference in mean change scores between week 2 and week 1 (scores for day 17 to day 10-scores for day 7 to day 1).
  Appetite loss was converted to a 0 til 100 scale according to the scoring manual for EORTC QLQ C15-PAL where 100 indicated maximum appetite loss (worst possible).
  Note outcome reported for complete compliers
Time Frame: One week
Population: Complete compliers
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Melatonin Then Placebo | Placebo Then Melatonin
Number analyzed (Participants) | 21 | 23
units on a scale | -0.8 (25.4) | -3.2 (21.6)

7. Secondary Outcome: General Fatigue Measured by the The Multidimensional Fatigue Inventory (MFI)
Description: Change from baseline to week one in intervention group minus change from baseline to week one in control group.
  Because it was a cross-over trial this was calculated the following way:
  Outcomes for arm 1 (melatonin then placebo) were calculated as the difference in mean change scores between week 1 and week 2 (scores for day 7 to day 1-scores for day 17 to day 10). Outcomes for arm 2 (placebo then melatonin) were calculated as the difference in mean change scores between week 2 and week 1 (scores for day 17 to day 10-scores for day 7 to day 1).
  The general fatigue scale that consits of four items was converted to a 0 til 100 scale where 100 indicated maximum (worst possible) fatigue.
  Note outcome reported for complete compliers
Time Frame: One week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Melatonin Then Placebo | Placebo Then Melatonin
Number analyzed (Participants) | 21 | 23
units on a scale | -3.2 (18.6) | -2.1 (24.8)

ADVERSE EVENTS:
Time Frame: SUSARS were registered for part 1 (two weeks plus washout phase) and part 2 (six weeks)
Description: Only SUSAR (suspected unexpected serious adverse reactions) are reported because the study population was patients in palliative care with many potential adverse events
  Data are not presented per intervention and since there were '0' SUSAR in both groups this does not matter.
Groups:
- Melatonin Then Placebo: Melatonin 20 mg melatonin orally every evening about 1 hour before bedtime for one week. Then placebo for one week.
- Placebo Then Melatonin: Placebo tablet orally every evening about one hour before bedtime for one week. Then melatonin 20 mg. for one week.
Arm/Group | Melatonin Then Placebo | Placebo Then Melatonin
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/38
Other Adverse Events (participants affected / at risk) | 0/34 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No